CLINICAL TRIAL: NCT05386810
Title: A Clinical Trial With an Open-label Phase to Evaluate the Safety of Five-dose Sabin Inactivated Poliovirus Vaccine (Vero Cell)（ msIPV） in Adults, Children and Infants, and a Blinded,Randomized and Controlled Phase to Evaluate the Lot Consistency Immunogenicity, and Safety of the msIPV in 2 Months Old Infants
Brief Title: Safety of Sabin Inactivated Poliovirus Vaccine in Adults, Children and Infants and Lot Consistency Immunogenicity, and Safety of the msIPV in 2 Months Old Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-msIPV-3001
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2022-05

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The clinical trial is divided into two stages: the first stage is an open design, and the second stage is a randomized ,blind control design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Safety group in adults (Experimental): 24 adults will receive one dose of 5-person sIPV vaccine to evaluate the safety of msIPV vaccine.
  Interventions: Biological: Experimental vaccine
- Safety group in children (Experimental): 24 children will receive one dose of 5-person sIPV vaccine to evaluate the safety of msIPV vaccine.
  Interventions: Biological: Experimental vaccine
- Safety group in infants (Experimental): 24 infants will receive 4 doses of vaccine according to the primary immunization schedule of 0,1,2 months and booster immunization schedule of 18 months to evaluate the safety of msIPV vaccine .
  Interventions: Biological: Experimental vaccine
- Experimental Vaccine-lot 1 (Experimental): 300 infants will receive 4 doses of 5-person sIPV vaccine of commercial scale lot 1 according to the primary immunization schedule of 0,1,2 months and booster immunization schedule of 18 months.
  Interventions: Biological: Experimental vaccine
- Experimental Vaccine-lot 2 (Experimental): 300 infants will receive 4 doses of 5-person sIPV vaccine of commercial scale lot 2 according to the primary immunization schedule of 0,1,2 months and booster immunization schedule of 18 months.
  Interventions: Biological: Experimental vaccine
- Experimental Vaccine-lot 3 (Experimental): 300 infants will receive 4 doses of 5-person sIPV vaccine of commercial scale lot 3 according to the primary immunization schedule of 0,1,2 months and booster immunization schedule of 18 months.
  Interventions: Biological: Experimental vaccine
- IPV control group (Active Comparator): 300 infants will receive 4 doses of IPV vaccine produced by Pasteur according to the primary immunization schedule of 0,1,2 months and booster immunization schedule of 18 months.
  Interventions: Biological: IPV control vaccine
- single-person sIPV control group (Active Comparator): 300 infants will receive 4 doses of single-dose sIPV vaccine produced by Pasteur according to the primary immunization schedule of 0,1,2 months and booster immunization schedule of 18 months.
  Interventions: Biological: single-person sIPV control vaccine

INTERVENTIONS:
Biological: Experimental vaccine — Sabin Inactivated Poliovirus Vaccine (Vero cell) (2.5ml)-investigational vaccine produced by Sinovac Biotech Co., Ltd. Inactivated Sabin poliovirus antigen (per 0.5ml): type 1 (15DU), type 2 (45DU), and type 3 (45DU)in 2.5 ml mixture of medium 199,glycine,formaldehyde,sodium chloride,potassium chloride,calcium chloride,magnesium sulfate,disodium phosphate,sodium dihydrogen phosphate,2 - phenoxyethanol for per injection.
  Other Names: msIPV
  Arms: Experimental Vaccine-lot 1; Experimental Vaccine-lot 2; Experimental Vaccine-lot 3; Safety group in adults; Safety group in children; Safety group in infants
Biological: IPV control vaccine — Inactivated Poliovirus Vaccine - control vaccine produced by Sanofi. Inactivated poliovirus antigens: Mahoney strain for type 1 (40DU), MEF-1 strain for type 2 (8DU), Saukett strains for type 3 (32DU) in 0.5 ml mixture of 2- phenoxyethanol,ethanol,formaldehyde,hanks199 medium (containing amino acids, mineral salts, vitamins, glucose, polysorbate 80 and water for injection),hydrochloric acid or sodium hydroxide (for pH value adjustment),trace amounts of antibiotics (neomycin, streptomycin and polymyxin B)for per injection.
  Arms: IPV control group
Biological: single-person sIPV control vaccine — Sabin Inactivated Poliovirus Vaccine (Vero cell) (0.5ml) -control vaccine produced by Sinovac Biotech Co., Ltd.
  Inactivated Sabin poliovirus antigen: type 1 (15DU), type 2 (45DU), and type 3 (45DU)in 0.5 ml mixture of medium 199,glycine,formaldehyde,sodium chloride,potassium chloride,calcium chloride,magnesium sulfate,disodium phosphate,sodium dihydrogen phosphate for per injection.
  Arms: single-person sIPV control group

SUMMARY:
This study includes two parts.A clinical trial with a open-label to evaluate the safety of Sabin Inactivated Poliovirus Vaccine (Vero cell) (2.5ml-5 doses)(hereinafter referred to as "msIPV")manufactured by Sinovac Biotech Co., Ltd. in adults, children and infants in partⅠ and a blinded,randomized and controlled clinical trial to evaluate the lot consistency immunogenicity, and safety of the msIPV in 2 months old infants in partⅡ.

DETAILED DESCRIPTION:
This study includes two stages. A clinical trial with an open-label to evaluate the safety of Sabin Inactivated Poliovirus Vaccine (Vero cell) (2.5ml-5 doses) (hereinafter referred to as "msIPV") in adults, children and infants in stageⅠ and a blinded, randomized and controlled clinical trial to evaluate the lot consistency immunogenicity, and safety of the msIPV in 2 months old infants in stage Ⅱ. A total of 1572 subjects including 24 adults aged 18-49 years,24 children aged 4 years,1524 infants aged 2 months will be enrolled.

StagesⅠ:72 healthy subjects, including 24 adults,24 children and 24 infants will be enrolled. 24 adults and 24 children will receive one dose of vaccine and 24 infants will receive 4 doses of vaccine according to the primary immunization schedule of 0,1,2 months and booster immunization schedule of 18 months.

StagesⅡ:1500 infants aged 2 months will be randomly divided into 5 groups (Experimental Vaccine-lot 1, Experimental Vaccine-lot 2, Experimental Vaccine-lot 3,IPV control group and single-dose sIPV control group) according to the ratio of 1:1:1:1:1. Subjects in 3 experimental groups will receive 5-dose sIPV produced by Sinovac for three lots, subjects in IPV control group will receive IPV produced by Pasteur, and subjects in single-dose sIPV control group will receive single-dose sIPV produced by Sinovac. All subjects will receive 4 doses of experimental or control vaccine according to the primary immunization schedule of 0,1,2 months, one dose of booster at 18 months of age.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for adult subjects :

* Healthy adults aged 18-49 days;
* Proven legal identification;
* The subject can understand and voluntarily sign the informed consent form.

Inclusion criteria for children subjects :

* Healthy children aged 4 years old;
* Subjects who have completed primary immunization with 3 doses of sIPV vaccine;
* Proven legal identification and vaccination certificate;
* The subject and/or guardian can understand and voluntarily sign the informed consent form.

Inclusion criteria for infant subjects:

* Healthy infants aged 2 months (60~89 days)
* Proven legal identification and vaccination certificate;
* The subject and/or guardian can understand and voluntarily sign the informed consent form.

Exclusion Criteria:

Exclusion criteria for adult subjects:

* Women aged 18 to 49 years, positive urine pregnancy test, pregnant women, breastfeeding women, or planning to become pregnant within 3 months;
* Previous history of vaccination of sIPV vaccine;
* Allergy history, history of asthma, including allergy history to vaccine or vaccine components, serious adverse reactions to the vaccine, such as urticaria, dyspnea, angioneurotic edema or stomachache, etc;
* Congenital malformation or developmental disorder, genetic defect, serious malnutrition, etc.;
* Autoimmune disease or immunodeficiency/immunosuppression;
* Thyroid disease or thyroidectomy history, absence of spleen, functional absence of spleen, and any conditions resulting in absence of spleen or splenectomy;
* Serious chronic diseases, serious cardiovascular diseases, hypertension that cannot be controlled by drugs (systolic blood pressure > 140mmHg, diastolic blood pressure > 90mmHg), diabetes, liver and kidney diseases, malignant tumors, etc;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Medical diagnosis of coagulation abnormalities (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities) or marked bruising or coagulation disorders;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids(excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* History of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Acute diseases or acute exacerbation of chronic diseases in the past 7 days;
* Axillary temperature >37.0°C;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Exclusion criteria for children subjects:

* Have received 4 doses of sIPV vaccine;
* History of polio;
* Allergy history, history of asthma, including allergy history to vaccine or vaccine components, serious adverse reactions to the vaccine, such as urticaria, dyspnea, angioneurotic edema or stomachache, etc;
* Congenital malformation or developmental disorder, genetic defect, serious malnutrition, etc.;
* Autoimmune disease or immunodeficiency/immunosuppression;
* Thyroid disease or thyroidectomy history, absence of spleen, functional absence of spleen, and any conditions resulting in absence of spleen or splenectomy;
* Suffering from serious cardiovascular diseases, diabetes, liver and kidney diseases, malignant tumors, etc;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Medical diagnosis of coagulation abnormalities (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities) or marked bruising or coagulation disorders;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids(excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* History of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Acute diseases or acute exacerbation of chronic diseases in the past 7 days;
* Axillary temperature >37.0°C;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Exclusion criteria for infant subjects:

* Previous history of vaccination of sIPV vaccine;
* History of polio;
* Allergy history, history of asthma, including allergy history to vaccine or vaccine components, serious adverse reactions to the vaccine, such as urticaria, dyspnea, angioneurotic edema or stomachache, etc;
* Preterm birth babies (delivered before 37 weeks gestation), low birth weight (girls with birth weight <2300g, boy with birth weight<2500 g);
* History of dystocia, asphyxia and nervous system damage at birth;

  * Congenital malformation or developmental disorder, genetic defect, serious malnutrition, etc.;
* Autoimmune disease or immunodeficiency/immunosuppression;
* Thyroid disease or thyroidectomy history, absence of spleen, functional absence of spleen, and any conditions resulting in absence of spleen or splenectomy;
* -Suffering from serious cardiovascular diseases, diabetes, liver and kidney diseases, malignant tumors, etc;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Medical diagnosis of coagulation abnormalities (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities) or marked bruising or coagulation disorders;
* Have received immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids(excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy);
* Receipt of blood products ;

  * Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Acute diseases or acute exacerbation of chronic diseases in the past 7 days;
* Axillary temperature >37.0°C;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 2 Months to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1572 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-10-08 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Safety index-incidence of adverse reactions | Within 30 days after each dose
  Incidence of adverse reactions within 30 days after each dose
Immunogenicity index-Geometric mean titers (GMT) | 30 days after primary immunization
  GMT 30 days after primary immunization in msIPV vaccination group
Immunogenicity index- seroconversion rate of neutralizing antibody | 30 days after primary immunization
  Seroconversion rate of neutralizing antibody 30 days after primary immunization in combined experiment group and IPV control group

SECONDARY OUTCOMES:
Safety index-incidence of adverse reactions | Within 7 days after each dose
  Incidence of adverse reactions within 7 days after each dose
Safety index-the incidence of adverse reactions | During the period of safety monitoring
  Incidence of SAE during the period of safety monitoring
Immunogenicity index- Neutralizing antibody positive rate and GMI | 30 days after primary immunization
  Neutralizing antibody positive rate and GMI and percentage of subjects with antibody ≥1:64 30 days after primary immunization
Immunogenicity index- Neutralizing antibody positive rate | Before booster dose
  Neutralizing antibody positive rate, percentage of subjects with antibody ≥1:64 and GMT before booster dose
Immunogenicity index-Neutralizing antibody positive rate,GMT and GMI | 30 days after booster dose
  Neutralizing antibody positive rate, percentage of subjects with antibody ≥1:64, GMT and GMI 30 days after booster dose

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Wang, Master, Principal Investigator — Henan Provincial Center for Disease Prevention and Control
Locations (2):
- China (2):
  - Xiangfu District Center for Disease Prevention and Control, Kaifeng, Henan
  - Xiangcheng County Center for Disease Control and Prevention, Xuchang, Henan